CLINICAL TRIAL: NCT04458246
Title: Online, Home-based, Aerobic Training Program Among Adolescents With Chronic Diseases During COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Home-based Aerobic Training Among Adolescents With Chronic Diseases During COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31314220.5.0000.0068
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Chronic Disease; Chronic Diseases in Adolescence; Chronic Disease of Immune System; Chronic Kidney Diseases
MeSH Terms: conditions — Chronic Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 10 patients from each chronic diseases conditions (1- Inflammatory bowel disease; 2- autoimmune hepatitis; 3- liver transplant; 4- renal transplant; 5- systemic lupus erythematosus; 6- juvenile dermatomyositis; 7- juvenile idiopathic arthritis) will receive an online home-based aerobic training, three times a week, during 3 months.
  Interventions: Other: Exercise training group
- Control (No Intervention): 10 patients from each chronic diseases conditions (1- Inflammatory bowel disease; 2- autoimmune hepatitis; 3- liver transplant; 4- renal transplant; 5- systemic lupus erythematosus; 6- juvenile dermatomyositis; 7- juvenile idiopathic arthritis) will be advised to maintain their daily routine.

INTERVENTIONS:
Other: Exercise training group — Online aerobic home-based exercise training, 3 times per week, during 3 months. The exercise program is composed by 3 levels (starter, intermediate and advanced) which be completed in the first, second and third month of intervention, respectively.
  Arms: Intervention

SUMMARY:
Data show that the coronavirus disease 2019 (COVID-19) symptoms can be severe in 4% and 3% of the adolescents aged 11-15 years and ≥ 16 years, respectively. In addition, the prevalence of chronic diseases among adolescents has increased in the last years. About 20% of the adolescents have some chronic disease, resulting in increased morbidity and mortality. In march, 2020, the quarantine was officially implemented in Sao Paulo, while elective medical appointments for adolescents with chronic disease were temporarily suspended. To mitigate the deleterious effect of the social isolation on physical and mental health among these patients, this study aims to test the effects of an online, home-based, exercise training program.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with either one of the following chronic conditions:

* Inflammatory bowel disease;
* autoimmune hepatitis;
* liver transplant;
* renal transplant;
* systemic lupus erythematosus;
* juvenile dermatomyositis;
* juvenile idiopathic arthritis.

Exclusion Criteria:

* Patients with physical limitations that preclude exercise.
* Patients diagnosed with COVID-19.
* Patients diagnosed with mental disorders.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of a home-based exercise training program | From baseline to 3 months of follow-up
  Semi structured interview

SECONDARY OUTCOMES:
Patients perceptions during social isolation | From baseline to 3 months of follow-up
  Semi structured interview
Adolescents quality of life | From baseline to 3 months of follow-up
  Quality of life will be assessed by means of Pediatric Quality of Life inventory (PedsQLTM 4.0)
Disease activity | From baseline to 3 months of follow-up
  Will be assessed by means of a visual analog scale (from 0 - no disease activity) to 10 - maximum disease activity).
Disease overall assessment | From baseline to 3 months of follow-up
  Will be assessed using the visual analog scale from 0 (very good condition) to 10 (very poor condition).
Strengths and difficulties | From baseline to 3 months of follow-up
  Will be assessed by means of Strengths & Difficulties Questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Univsersity of Sao Paulo, São Paulo, Brazil